CLINICAL TRIAL: NCT02013453
Title: A Phase II Randomized Trial Evaluating the Use of Proton Pump Inhibitors (PPIs) in Conjunction With Chemotherapy, in Patients With Recurrent Unresectable or Metastatic Cancers of the Head and Neck
Brief Title: A Phase II Trial of Proton Pump Inhibitors With Chemotherapy in Patients With Metastatic Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMCC 2013.046; HUM00074951 (Other: University of Michigan)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Omeprazole; Carboplatin; Fluorouracil; Paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observational (Active Comparator): Patients on the Observational arm are currently being treated with a proton pump inhibitor (PPIs) such as Omeprazole. They will receive standard of care chemotherapy. Standard treatment is the choice of the treating physician and may include Carboplatin in combination with either 5FU, Paclitaxel, or Pemetrexed.
  Interventions: Drug: Omeprazole; Drug: Carboplatin; Drug: 5FU; Drug: Paclitaxel; Drug: Pemetrexed
- Standard Chemo + Placebo (Active Comparator): Patients on the Standard Chemo and Placebo arm are not currently being treated with a proton pump inhibitor (PPI). They will be randomized to receive placebo along with standard of care chemotherapy. Standard treatment is the choice of the treating physician and may include Carboplatin in combination with either 5FU, Paclitaxel, or Pemetrexed.
  Interventions: Drug: Carboplatin; Drug: 5FU; Drug: Paclitaxel; Drug: Pemetrexed
- Standard Chemo + Omeprazole (Experimental): Patients on the Standard Chemo and Placebo arm are not currently being treated with a proton pump inhibitor (PPI). They will be randomized to receive Omeprazole along with standard of care chemotherapy. Standard treatment is the choice of the treating physician and may include Carboplatin in combination with either 5FU, Paclitaxel, or Pemetrexed.
  Interventions: Drug: Omeprazole; Drug: Carboplatin; Drug: 5FU; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Omeprazole — 40mg of Omeprazole will be administered daily by mouth.
  Arms: Observational; Standard Chemo + Omeprazole
Drug: Carboplatin — Carboplatin will be administered over 30 minutes by continuous infusion.
Drug: 5FU — Administered by infusion.
  Other Names: 5-Fluorouracil, Efudex
Drug: Paclitaxel — Administered by infusion.
Drug: Pemetrexed — Administered by infusion.

SUMMARY:
The purpose of this study is to determine if the addition of proton pump inhibitors (PPIs) to standard chemotherapy can improve progression free survival in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females at least 18 years old.
* Histologically or cytologically confirmed diagnosis of SCCHN (Squamous Cell Carcinoma of the Head and Neck).
* Stage IVC (metastatic) or advanced, locally recurrent SCCHN not amenable to curative surgery or radiotherapy.
* Measurable disease as defined by RECIST (Response Evaluation Criteria in Solid Tumors) vs 1.1 (Appendix 1).

  a. If the only site of measurable disease for this study is within a prior field of irradiation, then the sum of the longest diameters (SLD) of that lesion must have increased by at least 20% from the prior treatment nadir.
* ECOG Performance status (measure of health and general well being on a scale of 0 to 5 where 0 represents perfect health) < 1 (Appendix 2).
* Expected survival of at least 3 months.
* Adequate liver and renal function that is defined as Calculated creatinine clearance of <30ml/min (by Jelliffe calculator) AST (aspartate aminotransferase)/ALT (alanine aminotransferase) < 2.5 X ULN (unless there are hepatic metastasis, in which case AST/ALT within 5 X ULN) Total Bilirubin < 1.5 X ULN (Appendix 5).
* Ability to understand and willingness to sign an informed consent form.
* Willingness and ability to comply with study procedures and follow up.
* There is no restriction on number of prior therapies as long as the patient is deemed a candidate for palliative chemotherapy with one of the standard chemotherapy regimens.
* Willingness to use contraception by a method that is deemed effective by the Investigator by both male and female patients of childbearing potential and their partners throughout the treatment period and for at least 30 days following the last cycle of chemotherapy (post menopausal women must have been amenorrheal for at-least 12 months to be considered of non-childbearing potential).

Exclusion Criteria:

* Comorbidities precluding treatment with combination chemotherapy or per investigator discretion.
* Pregnancy or lactation.
* Medical or psychiatric illness that may compromise the patient's ability to tolerate the treatment or comply with the study requirements.
* Patients with another active cancer or history of another cancer in the last 3 years except those treated with curative intent such as skin cancer (other than melanoma), in situ breast or in situ cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
* Allergy to PPI or inability to tolerate PPI.
* Patients residing in prison.
* Any investigational drug dose within 28 days of planned start of trial.
* Any concurrent standard therapy intended to treat SCCHN.
* Any symptomatic infection (bacterial, fungal or viral) as per the investigator discretion.
* Patients with uncontrolled CNS (Central Nervous System) metastases are excluded. Patients with known, previously treated CNS metastases are eligible if they are neurologically stable as per the investigating physician's clinical assessment.
* Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
* Patients on Rilpivirine, Atazanavir, Indinavir and Nelfinavir will not be eligible for participation in study because of the significant drug interaction unless the patient can be switched to a different antiviral medication prior to study enrollment.
* Omeprazole can increase the serum concentration of methotrexate, clorazepate and citalopram increasing the risk of adverse effects.
* Omeprazole may result in reduction in clinical efficacy of clopidogrel and increased risk for thrombosis.
* Omeprazole when co-administered with dasatinib, bosutinib, ponatinib, erlotinib, dabrafenib and vismodegib reduces the systemic exposure to these drugs, therefore patients on these drugs should not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 6 months post treatment
  The primary aim, progression-free survival, will be defined from start of treatment to date of first progression and will be tested using a Cox proportional hazard regression model with treatment arm as the only predictor.

SECONDARY OUTCOMES:
Median overall survival | 6 months post treatment
  Overall survival be evaluated with Cox models and will be defined from the first date of treatment to date of death.
Proportion of patients that experience a response to treatment | 6 months post treatment
  Estimate the proportion of patients with a complete response (CR), partial response (PR), objective response (CR+PR) and clinical benefit (CR+PR+Stable disease) and compare responses between the group receiving proton pump inhibitors (PPI) and the group not receiving PPIs.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States